CLINICAL TRIAL: NCT07248982
Title: Prospective Cohort Study of High-Strength Suture Modified Tension Band Technique for the Treatment of Patellar Fractures
Brief Title: High-Strength Suture vs. Traditional Tension Band for Patellar Fractures
Status: Recruiting | Type: Observational
Sponsor: Fuzhou University Affiliated Provincial Hospital (Other)
Responsible Party: Principal Investigator, Anning Liu, Anning Liu, Emergency Medicine Graduate, Fujian medical university, Fuzhou University Affiliated Provincial Hospital
Other Study IDs: K2025-10-005
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Patella Fracture
Keywords: Patellar Fracture; Tension Band Fixation; High-Strength Suture; Knee Function; Lysholm Score; VAS Pain Score; Prospective Cohort
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suture Fixation (SF) Group: Patients receiving high-strength suture modified tension band fixation for patellar fracture.
  Interventions: Procedure: High-Strength Suture Modified Tension Band Fixation
- Screw-Cable Tension Band (SCTB) Group: Patients receiving traditional screw-cable tension band fixation for patellar fracture.
  Interventions: Procedure: Screw-Cable Tension Band Fixation

INTERVENTIONS:
Procedure: High-Strength Suture Modified Tension Band Fixation — Use of high-strength sutures for modified tension band fixation in patellar fracture surgery.
  Other Names: Suture Fixation (SF)
  Groups: Suture Fixation (SF) Group
Procedure: Screw-Cable Tension Band Fixation — Use of screws and cables for traditional modified tension band fixation in patellar fracture surgery.
  Groups: Screw-Cable Tension Band (SCTB) Group

SUMMARY:
This prospective cohort study aims to evaluate the clinical efficacy of high-strength suture modified tension band fixation in treating patellar fractures and compare it with traditional screw-cable tension band fixation. Adult patients (18-55 years) with AO/OTA 34-C1 or 34-C2 patellar fractures will be enrolled and followed for 12 months. Primary outcomes include Lysholm knee function score, knee range of motion (ROM), and visual analog scale (VAS) pain score at 12 months post-surgery. Secondary outcomes include fracture healing time, radiographic alignment quality, complication rates, reoperation rates, implant removal rates, SF-36 health survey scores, and patient satisfaction. No additional biological samples will be collected; data will focus on clinical, radiographic, and follow-up information.

DETAILED DESCRIPTION:
Patellar fractures account for approximately 1% of all fractures and are common in knee injuries. Traditional tension band fixation is widely used but associated with issues such as hardware migration, soft tissue irritation, and postoperative pain, impacting rehabilitation and quality of life. High-strength sutures offer improved biomechanical properties, flexibility, and reduced soft tissue damage. This study observes the clinical efficacy of high-strength suture modified tension band fixation compared to traditional methods through a prospective cohort design.

Patients admitted to Fuzhou University Affiliated Provincial Hospital from February 2024 to February 2026 with patellar fractures undergoing surgery will be divided into two groups based on surgical method: Suture Fixation (SF) group and Screw-Cable Tension Band (SCTB) group. Follow-up will occur for 12 months, assessing outcomes such as postoperative VAS pain scores, Lysholm knee scores, ROM, SF-36 health surveys, surgical time, intraoperative blood loss, hospital stay, and complications (e.g., infection, fixation failure, nonunion).

General data collected includes demographics (age, gender, height, weight, BMI), comorbidities (e.g., diabetes, hypertension, smoking), ASA classification, fracture details (side, type, displacement, mechanism, time from injury), and perioperative complications. Imaging assessments include fracture reduction quality (good, satisfactory, poor) via X-ray, healing time (weeks until fracture line blurs/disappears), and patellar height via Insall-Salvati index. Muscle strength (quadriceps via MMT, 0-5 grades) and patient satisfaction (1-5 scale) will also be evaluated.

Adverse events (AEs) and serious adverse events (SAEs) will be recorded, reported to the ethics committee, and managed promptly. Statistical analysis will use IBM SPSS Statistics 27.0, with t-tests, Mann-Whitney U tests, chi-square/Fisher's exact tests, Kaplan-Meier curves, and regressions as appropriate. Intention-to-treat (ITT) analysis will be primary, with multiple imputation for missing data.

The study is feasible given the hospital's patient volume and the principal investigator's experience. Ethical principles follow the Helsinki Declaration, with informed consent and privacy protection. Results will be published in academic journals and presented at conferences.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-55 years. 2.Radiographically confirmed patellar fracture (AO/OTA 34-C1 or 34-C2). 3.First-time patellar fracture surgery. 4.Time from injury to surgery ≤ 2 weeks. 5.Able to comply with follow-up and provide written informed consent. 6.Normal pre-injury knee function. 7.Able to tolerate surgery and agree to surgical treatment. 8.Intact cognitive function.

Exclusion Criteria:

* 1.Age <18 or >55 years. 2.Pathological fractures. 3.Prior patellar surgery or severe underlying patellofemoral disease. 4.Time from injury to surgery >2 weeks. 5.Concurrent active infection or severe medical conditions. 6.Severe neuropsychiatric disorders affecting follow-up compliance. 7.Postmenopausal women. 8.Inability to tolerate surgery or refusal of surgery. 9.Comorbid patellar dysplasia, rheumatoid arthritis, or other patellofemoral diseases.

  10.Comorbid systemic or local infection at surgical site. 11.Comorbid severe lower limb or systemic injuries. 12.Pre-injury cognitive impairment, mental disorder, or independent walking disability.

  13.Other conditions unsuitable for enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with patellar fractures seeking surgical treatment at Fuzhou University Affiliated Provincial Hospital, meeting inclusion criteria, and grouped based on surgical technique received.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Score at 12 Months Postoperatively | 12 months postoperatively
  Lysholm knee scoring scale (0-100 points; 95-100 = excellent, 84-94 = good, 65-83 = fair, <65 = poor; higher scores indicate better knee function). Assessed at baseline (pre-injury recalled), 1 week, 1 month, 3 months, 6 months, and 12 months postoperatively.
Knee Range of Motion at 12 Months Postoperatively | 12 months postoperatively
  Active knee flexion and extension range of motion measured in degrees with a goniometer (higher values indicate better function). Assessed at 1 week, 1 month, 3 months, 6 months, and 12 months postoperatively.
Visual Analog Scale (VAS) Pain Score at 12 Months Postoperatively | 12 months postoperatively
  Visual Analog Scale for pain (0-10 points; 0 = no pain, 10 = worst imaginable pain; higher scores indicate more severe pain). Assessed preoperatively and at 1 week, 1 month, 3 months, 6 months, and 12 months postoperatively.

SECONDARY OUTCOMES:
Fracture Healing Time | Assessed at 6 weeks, 3 months, 6 months, and 12 months postoperatively or until healing confirmed
  Time in weeks from surgery until radiographic evidence of fracture line blurring or disappearance on X-ray/CT.
Radiographic Alignment Quality | Immediately postoperatively and at 1 month, 3 months, 6 months, and 12 months postoperatively
  Postoperative fracture reduction quality graded as good, satisfactory, or poor based on X-ray.
Complication Rate | From surgery to 12 months postoperatively
  Incidence of any postoperative complications (e.g., infection, fixation failure, nonunion, knee stiffness, deep vein thrombosis).
Reoperation Rate | From surgery to 12 months postoperatively
  Percentage of patients requiring any additional surgery related to the index fracture.
Implant Removal Rate | From surgery to 12 months postoperatively
  Percentage of patients requiring removal of surgical implants.
SF-36 (36-Item Short Form Health Survey) Score | 12 months postoperatively
  36-Item Short Form Health Survey (SF-36) questionnaire assessing health-related quality of life. The SF-36 includes eight domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health); scores for each domain range from 0-100, with higher scores indicating better health status. The Physical Component Summary (PCS) and Mental Component Summary (MCS) will also be calculated and reported. Assessed at 12 months postoperatively.
Surgical Time | Day of surgery
  Duration of the surgical procedure recorded in minutes from skin incision to closure.
Intraoperative Blood Loss | Day of surgery
  Estimated volume of blood loss during surgery recorded in milliliters.
Hospital Stay Duration | From day of surgery to discharge
  Number of days from the date of surgery to the date of hospital discharge.
Quadriceps Muscle Strength (Manual Muscle Testing) | Assessed at 1 week, 1 month, 3 months, 6 months, and 12 months postoperatively
  Quadriceps strength graded 0-5 using Manual Muscle Testing (MMT; 0 = no contraction, 5 = normal strength), compared with the contralateral side.
Patellar Height (Insall-Salvati Index) | Assessed at 1 month, 3 months, 6 months, and 12 months postoperatively
  Ratio of patellar tendon length to patellar length measured on lateral knee radiographs (normal range 0.8-1.2).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Dr, Principal Investigator — Fuzhou University Affiliated Provincial Hospital
Locations (1):
- Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated study results and summary statistics will be made available through publications and conference presentations.

REFERENCES:
- [Background] Adjal J, Haugaard A, Vesterby L, Ibrahim HM, Sert K, Thomsen MG, Tengberg PT, Ban I, Ohrt-Nissen S. Suture tension band fixation vs. metallic tension band wiring for patella fractures - A biomechanical study on 19 human cadaveric patellae. Injury. 2022 Aug;53(8):2749-2753. doi: 10.1016/j.injury.2022.05.015. Epub 2022 May 26. PMID 35701245
- [Background] Hughes SC, Stott PM, Hearnden AJ, Ripley LG. A new and effective tension-band braided polyester suture technique for transverse patellar fracture fixation. Injury. 2007 Feb;38(2):212-22. doi: 10.1016/j.injury.2006.07.013. Epub 2006 Nov 13. PMID 17098238
- [Background] Carpenter JE, Kasman RA, Patel N, Lee ML, Goldstein SA. Biomechanical evaluation of current patella fracture fixation techniques. J Orthop Trauma. 1997 Jul;11(5):351-6. doi: 10.1097/00005131-199707000-00009. PMID 9294799
- [Background] LeBrun CT, Langford JR, Sagi HC. Functional outcomes after operatively treated patella fractures. J Orthop Trauma. 2012 Jul;26(7):422-6. doi: 10.1097/BOT.0b013e318228c1a1. PMID 22183197
- [Background] Sayum Filho J, Lenza M, Tamaoki MJ, Matsunaga FT, Belloti JC. Interventions for treating fractures of the patella in adults. Cochrane Database Syst Rev. 2021 Feb 24;2(2):CD009651. doi: 10.1002/14651858.CD009651.pub3. PMID 33625743
- [Background] Huang L, Li X, Ye L, Li S. Closed Reduction and High-Strength Sutures for Transverse Patella Fractures: A Retrospective Analysis. Indian J Orthop. 2023 Feb 27;57(4):571-576. doi: 10.1007/s43465-023-00843-4. eCollection 2023 Apr. PMID 37006729
- [Background] Giuseppe R, Michele R, Luca F, Michele G, Giuseppe G, Valentina M, Giustra F, Bosco F, Camarda L. Nonmetallic tension band fixation is a viable and low-complication surgical technique in patellar fractures: a five-year retrospective study. Eur J Orthop Surg Traumatol. 2024 May;34(4):2065-2071. doi: 10.1007/s00590-024-03887-w. Epub 2024 Mar 26. PMID 38530504
- [Background] Xiang F, Xiao Y, Li D, Ma W, Chen Y, Yang Y. Tension band high-strength suture combined with absorbable cannulated screws for treating transverse patellar fractures: finite element analysis and clinical study. Front Bioeng Biotechnol. 2024 Mar 7;12:1340482. doi: 10.3389/fbioe.2024.1340482. eCollection 2024. PMID 38515618

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT07248982/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT07248982/ICF_001.pdf